CLINICAL TRIAL: NCT02558907
Title: Comparison of MMSE (Mini-Mental State Examination) and MoCA (Montreal Cognitive Assessment) in Cognitive Assessment in Geriatric Oncology
Acronym: MoCA
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: MoCA
Record Dates: First submitted 2015-09-18; First posted 2015-09-24 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2016-06

CONDITIONS: Geriatrics; Cancer
Keywords: geriatrics; cancer; MMS test; MoCA test; cognitive evaluation
MeSH Terms: conditions — Neoplasms | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cognitive evaluation by MMS (Mini-Mental State Examination) and MoCA (Montreal Cognitive Assessment) tests

SUMMARY:
Compare neurocognitive testing MMSE (Mini-Mental State Examination) and MoCA (Montreal Cognitive Assessment) to candidates aged patients with 1st line treatment of their cancer will be received an examination oncogériatric

ELIGIBILITY:
Inclusion Criteria:

* Patient old over 70 years
* Patient with cancer (solid tumor or hematological) for which a 1st line treatment is planned
* Patient candidate an oncogeriatric assessment
* Patient agreeing to participate in the study
* French language
* Lack of subsequent neurological sequelae with cognitive impact stroke, dementia or progressive psychiatric disorder
* Patient having a life expectancy ≥ 6 months

Exclusion Criteria:

* Primitive cancer of the central nervous system or brain metastasis
* Patients unable to meet the cognitive tests
* Refusal to participate
* Realization of a MMSE or MoCA test in the last 6 months

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: aged patients with 1st line treatment of their cancer will be received an examination oncogériatric
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
proportion of patients with cognitive disorders identified by the MoCA or the MMSE prior to treatment | before their first treatment for the cancer, at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Heidi LAVIEC, MD, Principal Investigator — Centre François Baclesse - CAEN
Locations (2):
- France (2):
  - CHU, Caen
  - Centre François Baclesse, Caen